CLINICAL TRIAL: NCT02505464
Title: Characteristics of Pregnancies Complicated by Fetal Anomalies
Brief Title: Pregnancies Complicated by Fetal Anomalies
Acronym: FAR
Status: Recruiting | Type: Observational
Sponsor: University of Tennessee (Other)
Collaborators: Regional One Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-03804-XP
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy; Congenital Abnormalities
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women & their fetuses/infants: Information about pregnant women and their fetuses/infants, including the medical history, prenatal, perinatal, and postpartum periods (6 weeks after delivery) and throughout the treatment (e.g.surgery) for the child's medical condition (up to approx. child is @ 6 months of age), will be collected in this repository. The analysis of this information may help in understanding of the causes of fetal anomalies.

SUMMARY:
The focus of this research is to create a repository of ultrasonographic images and their corresponding medical data from pregnant women (the mothers of the fetuses that are imaged), focusing on fetal anomalies. These women will visit the obstetrical clinics at Regional One Health and the Le Bonheur Fetal Center.

DETAILED DESCRIPTION:
1. Repository data will be collected from the medical record and entered into the data base after the patient has completed the appointment.
2. Data collection will continue into the postpartum period for each participant.
3. Data collection will continue for the child during the treatment of the medical condition, up to approximately 6 months of age if required by the condition.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females

  * age 8 years to 50 years
  * who have referred to the clinic for high risks pregnancies
* Infants (male and female) born with anomalies

Exclusion Criteria:

* Non-pregnant females.

Ages: 1 Minute to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients referred to, or being seen in the Ob-Gyn High Risk Clinics (ROH-MFM Clinic, ROH-CHRP, ROH-Rout Center, Le Bonheur Fetal Center) will be potential participants.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Data Collection | From the initial visit @ the High Risk Clinic through the infants approx. age of 6 months
  Data collection from participant's medical records will be entered into a data base

CONTACTS AND LOCATIONS:
Overall Officials: Norman Meyer, M.D., Principal Investigator — Vice-Chair and Professor, MFM Fellowship Director Obstetrics and Gynecology
Locations (5):
- United States (5):
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Methodist LeBonheur Healthcare, LeBonheur Fetal Center, Memphis, Tennessee
  - Regional One Health, OB/GYN Clinic, Maternal Fetal Medicine, Memphis, Tennessee
  - Regional One Health, Regional Medical Center, Rout Center for Women and Children, Memphis, Tennessee
  - Regional One Health Center for High Risk Pregnancies, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided